CLINICAL TRIAL: NCT05600881
Title: Understanding the Mechanism of Action of Methylphenidate in ADHD: A Computational Psychiatry Approach
Brief Title: Towards an Understanding of the Mechanism of Action of Methylphenidate in ADHD
Status: Not yet recruiting | Type: Observational
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Julia Paterson, PhD Candidate, University of Dublin, Trinity College
Other Study IDs: MPH2022TCD
Record Dates: First submitted 2022-10-26; First posted 2022-11-01 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ADHD: This study will recruit people aged 14-17 with ADHD who are 'Assigned Female At Birth' (AFAB). This is to include cisgender women alongside those who may not identify with womanhood such as those who are non-binary but AFAB or transgender men who have not undergone hormonal/medical transition.
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate — Participants will take their regular medication or a placebo (vitamin C)

SUMMARY:
Approximately 1-in-20 children worldwide have Attention Deficit Hyperactivity Disorder (ADHD), a condition associated with disabling inattention, hyperactivity and impulsivity. These problems can manifest as poor inhibitory control (e.g., difficulty holding back impulsive actions) and atypical reward processing (e.g., failing to learn from adverse outcomes). Poorly treated ADHD is associated with negative academic and socioeconomic consequences.

This project aims to ultimately improve clinical management of children with ADHD. Methylphenidate, a stimulant medication, is used as the first-option pharmacological treatment for ADHD and often successfully reduces problem behaviour. Although Methylphenidate can be extremely effective, it does not work for every child. There is currently no 'objective' way (e.g., blood test or brain scan) to measure if a child is genuinely responding to Methylphenidate. Instead, clinicians must rely on reports from parents and teachers, an approach that is problematic and that often leads to delays in optimising ADHD treatment. The absence of a biological test to quantify Methylphenidate response is primarily because we do not understand exactly how Methylphenidate changes behaviours to produce the known beneficial effects. This lack of knowledge is despite the very common use of this medication.

This project will investigate the specific brain processes that are affected by Methylphenidate by recording brain activity and behaviour in children with ADHD (who have already been prescribed Methylphenidate as part of their clinical care) when they are on and off this medication. Brain activity will be recorded using two separate approaches, which are both non-invasive and routinely used in Trinity College Institute of Neuroscience: electroencephalography (EEG) and functional magnetic resonance imaging (fMRI). Brain activity data will be collected while children with ADHD are performing two computer-game like tasks. One task measures the child's ability to hold back impulsive actions (inhibition) and the other assesses how they learn from positive and negative outcomes (reward processing). The data from the two tasks, the EEG recording and the fMRI scan will be analysed using advanced computer-modelling approaches to determine exactly how Methylphenidate changes behaviour.

This project is important because if we can understand the brain mechanisms affected by Methylphenidate, we can ultimately develop a computerised measure that will allow clinicians to predict whether a child is going to respond to this treatment or not. Such a measure would allow clinicians to treat ADHD more effectively and would result in children with ADHD experiencing faster relief from symptoms.

DETAILED DESCRIPTION:
This project will investigate the specific brain processes that are affected by Methylphenidate by recording brain activity and behaviour in children with ADHD (who have already been prescribed Methylphenidate as part of their clinical care) when they are on and off this medication.

This is a quantitative double-blind placebo-controlled study investigating the acute effects of methylphenidate on brain activity using two non-invasive methods, EEG and fMRI.

Brain activity will be recorded using two separate approaches, which are both non-invasive and routinely used in Trinity College Institute of Neuroscience: electroencephalography (EEG) and functional magnetic resonance imaging (fMRI). Brain activity data will be collected while children with ADHD are performing two computer-game like tasks. One task measures the child's ability to hold back impulsive actions (inhibition) and the other assesses how they learn from positive and negative outcomes (reward processing). The data from the two tasks, the EEG recording, and the fMRI scan will be analysed using advanced computer-modelling approaches to determine exactly how Methylphenidate changes behaviour.

ELIGIBILITY:
Inclusion Criteria:

AFAB Clinical diagnosis of ADHD Must be able to swallow tablets Regular menstrual cycles Good response to medication

Exclusion Criteria:

Intellectual Disability Specific Learning Disabilities

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Assigned Female At Birth (AFAB)
Study Population: Approximately 35 participants aged 14-17 years old will be recruited.
  As previous research on ADHD has overwhelmingly focussed on cisgender men, this study will recruit people who are 'Assigned Female At Birth' (AFAB). This is to include cisgender women alongside those who may not identify with womanhood such as those who are non-binary but AFAB or transgender men who have not undergone hormonal/medical transition.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
MRI | 2023-2026
  structural, diffusion, functional

SECONDARY OUTCOMES:
Stop Signal Task | 2023-2026
  behavioural measures

OTHER OUTCOMES:
EEG | 2023-2026
  during SST

IPD SHARING:
Plan to Share IPD: Undecided